CLINICAL TRIAL: NCT02213471
Title: Patient Preference for Biopsy Notification
Status: Completed | Type: Observational
Sponsor: Maria Wei (Other)
Responsible Party: Sponsor-Investigator, Maria Wei, Associate Professor of Dermatology, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Other Study IDs: BX001
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Elevated Risk for Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Elevated risk for melanoma: Individuals at increased risk for melanoma due to past history of melanoma, family history of melanoma, the presence of many moles, the presence of a genetic mutation known to increase the risk of melanoma.

SUMMARY:
Effective communication between physician and patient is fundamental to effective care. The recent introduction of electronic patient on-line portals has the potential to change the communication landscape. The investigators surveyed patients to assess their preferred modality for biopsy notification at 3 institutions with differing patient access to on-line portals, to ascertain what patient preferences are currently and if it has changed from historical preferences. Our hypothesis is that as patients become more familiar with ln-line portals, their preferences will likely reflect familiarity with this modality.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were 18 years of age or older and English speaking were eligible to participate

Exclusion Criteria:

* Younger than 18, non-English speaking.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals at increased risk for melanoma due to past history of melanoma, family history of melanoma, the presence of many moles, the presence of a genetic mutation known to increase the risk of melanoma. Individuals were followed in a Pigmented Lesion Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Patient preference for biopsy notification | 1 year
  Patients were asked to rank in order of preference their preferred method for being notified of a skin biopsy result

CONTACTS AND LOCATIONS:
Overall Officials: Maria L Wei, MD PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States